CLINICAL TRIAL: NCT01101841
Title: A Phase 3, Twenty-Four Week, Multicenter, Double-Blind, Randomized, Placebo-Controlled, Efficacy and Safety Study of Mesafem (Paroxetine Mesylate) Capsules in the Treatment of Vasomotor Symptoms Associated With Menopause
Brief Title: 24-Week Efficacy & Safety Study of Brisdelle™ (Formerly Known as Mesafem) in the Treatment of Vasomotor Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Noven Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N30-004
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Hot Flashes
Keywords: Vasomotor Symptoms; Menopause; Hot Flashes; Perimenopause; Nonhormonal therapies; Climacteric symptoms; Mesafem; Low-Dose Mesylate salt of Paroxetine (LDMP)
MeSH Terms: conditions — Hot Flashes | interventions — Paroxetine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brisdelle (paroxetine mesylate) (Experimental): Brisdelle (paroxetine mesylate)
  Interventions: Drug: Brisdelle (paroxetine mesylate)
- Placebo capsules (Placebo Comparator): Sugar pill
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: Brisdelle (paroxetine mesylate) — Eligible subjects will be randomized to receive either Brisdelle (paroxetine mesylate) Capsules 7.5 mg or placebo capsules in a 1:1 ratio.
  Other Names: Former Names: Mesafem Capsules or; LDMP (Low-Dose Mesylate salt of Paroxetine)
  Arms: Brisdelle (paroxetine mesylate)
Drug: Placebo capsules — Eligible subjects will be randomized to receive either Brisdelle (paroxetine mesylate) Capsules 7.5 mg or placebo capsules in a 1:1 ratio.
  Other Names: Sugar pill
  Arms: Placebo capsules

SUMMARY:
To assess the safety and efficacy of Brisdelle (paroxetine mesylate) Capsules 7.5 mg for treatment of vasomotor symptoms (VMS) associated with menopause

DETAILED DESCRIPTION:
The study is a 24-week, multicenter, double-blind, randomized, placebo-controlled study of Brisdelle (paroxetine mesylate) Capsules 7.5 mg in subjects with moderate to severe postmenopausal VMS, defined as follows:

1. Moderate VMS: Sensation of heat with sweating, able to continue activity
2. Severe VMS: Sensation of heat with sweating, causing cessation of activity

The study is comprised of a screening period, a run-in period, a baseline visit, and a double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Female, >40 years of age
2. Reported more than 7-8 moderate to severe hot flashes per day (average) or 50-60 moderate to severe hot flashes per week for at least 30 days prior
3. Spontaneous amenorrhea for at least 12 consecutive months
4. Amenorrhea for at least 6 months and meet the biochemical criteria for menopause
5. Bilateral salpingo-oophorectomy >6 weeks with or without hysterectomy

Exclusion Criteria:

1. BMI ≥ 40 kg/m²
2. Known non-responder to previous Selective serotonin reuptake inhibitor (SSRI) or Serotonin norepinephrine reuptake inhibitor (SNRI) treatment for VMS
3. History of self-injurious behavior
4. History of clinical diagnosis of depression; or treatment for depression
5. History of clinical diagnosis of borderline personality disorder
6. Use of an investigational study medication within 30 days prior to screening or during the study
7. Concurrent participation in another clinical trial or previous participation in this trial
8. Family of investigational-site staff

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2010-03; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derrick R Havin, MD, Principal Investigator — North Spokane Women's Clinic Research, Spokane, WA 99207; Richard E Hedrick, MD, Principal Investigator — Hawthorne Medical Research, Inc., Winston-Salem, NC 27103; Samuel N Lederman, MD, Principal Investigator — Altus Research, Lake Worth, FL 33461; Larry S Seidman, DO, Principal Investigator — Philadelphia Clinical Research, LLC, Philadelphia, PA 19114; James E Tomblin, MD, Principal Investigator — Hawthorne Medical Research, Inc., Greensboro, NC 27408; Peter A Zedler, MD, Principal Investigator — Virginia Women's Center, Richmond, VA 23233; D S Harnsberger, MD, Principal Investigator — Chattanooga Medical Research, LLC, Chattanooga, TN 37404; John A Hoekstra, MD, Principal Investigator — National Clinical Research, Inc., Richmond, VA 23294; Robin Kroll, MD, Principal Investigator — Women's Clinical Research Center, Seattle, WA 98105; Ashley Tunkle, MD, Principal Investigator — Anchor Research Center, Naples, FL 34102; Matthew Davis, MD, Principal Investigator — Rochester Clinical Research, Rochester, NY 14609; Donna DeSantis, MD, Principal Investigator — East Valley Family Physicians PLC, Chandler, AZ 85224; Steven Drosman, Principal Investigator — Genesis Center For Clinical Research, San Diego, CA 92103; Mildred Farmer, MD, Principal Investigator — Meridien Research, Brooksville, FL 34601; Sandra Hurtado, MD, Principal Investigator — The Woman's Hospital of Texas Clinical Research Center, Houston, TX 77054; Bruce Levine, MD, Principal Investigator — Phoenix Ob-Gyn Associates, LLC, Moorestown, NJ 08057; Tyrone Malloy, MD, Principal Investigator — Soapstone Center for Clinical Research, Decatur, GA 30034; Eric Ross, MD, Principal Investigator — Apex Research Institute, Santa Ana, CA 92705; Cynthia Strout, MD, Principal Investigator — Coastal Carolina Research Center, Mt. Pleasant, SC 29464; Arthur Waldbaum, MD, Principal Investigator — Downtown Women's Health Care, Denver, CO, 80218; Edward Zbella, MD, Principal Investigator — Women's Medical Research Group, LLC, Clearwater, FL 33759; James R Dockery, MD, Principal Investigator — Montgomery Women's Health Associates, PC, Montgomery, AL 36116; Stephen C Blank, MD, Principal Investigator — Mount Vernon Clinical Research, LLC, Sandy Springs, GA 30328; Keith Aqua, MD, Principal Investigator — Visions Clinical Research, Boynton Beach, FL 33472; Saul R Berg, MD, Principal Investigator — Clinical Trials Research Services, LLC, Pittsburgh, PA 15206; Marvin Kalafer, MD, Principal Investigator — The Clinical Trial Center, LLC, Jenkintown, PA 19046; David J Portman, MD, Principal Investigator — Columbus Center for Women's Health Research, Columbus, Ohio 43213; Stephen Swanson, MD, Principal Investigator — Women's Clinic of Lincoln, PC, Lincoln, NE 68510; Joseph Soufer, MD, Principal Investigator — Chase Medical Research, LLC, Waterbury, CT 06708; ShaH R Scott, MD, Principal Investigator — Clinical Research Associates, Inc., Nashville, TN 37203; Mary K Neuffer, MD, Principal Investigator — SC Clinical Research Center, LLC, Columbia, SC 29201; Ronald Ackerman, MD, Principal Investigator — Comprehensive Clinical Trials, LLC, West Palm Beach, FL 33409
Locations (32):
- United States (32):
  - Montgomery Women's Health Associates, PC, Montgomery, Alabama
  - East Valley Family Physicians PLC, Chandler, Arizona
  - Genesis Center For Clinical Research, San Diego, California
  - Apex Research Institute, Santa Ana, California
  - Downtown Women's Health Care, Denver, Colorado
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Visions Clinical Research, Boynton Beach, Florida
  - Meridien Research, Brooksville, Florida
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Altus Research, Lake Worth, Florida
  - Anchor Research Center, Naples, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Soapstone Center for Clinical Research, Decatur, Georgia
  - Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Women's Clinic of Lincoln, PC, Lincoln, Nebraska
  - Phoenix Ob-Gyn Associates, LLC, Moorestown, New Jersey
  - Rochester Clinical Research, Rochester, New York
  - Hawthorne Research, Greensboro, North Carolina
  - Hawthorne Medical Research, Inc., Winston-Salem, North Carolina
  - Columbus Center for Women's Health Research, Columbus, Ohio
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Philadelphia Clinical Research, Philadelphia, Pennsylvania
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - SC Clinical Research Center, LLC, Columbia, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - The Woman's Hospital of Texas Clinical Research Center, Houston, Texas
  - Virginia Women's Center, Richmond, Virginia
  - National Clinical Research, Inc., Richmond, Virginia
  - Women's Clinical Research Center, Seattle, Washington
  - North Spokane Women's Clinic Research, Spokane, Washington

REFERENCES:
- [Background] Fugate SE, Church CO. Nonestrogen treatment modalities for vasomotor symptoms associated with menopause. Ann Pharmacother. 2004 Sep;38(9):1482-99. doi: 10.1345/aph.1D610. Epub 2004 Aug 3. PMID 15292498
- [Background] Kritz-Silverstein D, Goldani Von Muhlen D, Barrett-Connor E. Prevalence and clustering of menopausal symptoms in older women by hysterectomy and oophorectomy status. J Womens Health Gend Based Med. 2000 Sep;9(7):747-55. doi: 10.1089/15246090050147727. PMID 11025867
- [Background] Nelson HD, Vesco KK, Haney E, Fu R, Nedrow A, Miller J, Nicolaidis C, Walker M, Humphrey L. Nonhormonal therapies for menopausal hot flashes: systematic review and meta-analysis. JAMA. 2006 May 3;295(17):2057-71. doi: 10.1001/jama.295.17.2057. PMID 16670414
- [Background] Greene JG. A factor analytic study of climacteric symptoms. J Psychosom Res. 1976;20(5):425-30. doi: 10.1016/0022-3999(76)90005-2. No abstract available. PMID 1003364
- [Derived] Pinkerton JV, Joffe H, Kazempour K, Mekonnen H, Bhaskar S, Lippman J. Low-dose paroxetine (7.5 mg) improves sleep in women with vasomotor symptoms associated with menopause. Menopause. 2015 Jan;22(1):50-8. doi: 10.1097/GME.0000000000000311. PMID 25137243
- [Derived] Portman DJ, Kaunitz AM, Kazempour K, Mekonnen H, Bhaskar S, Lippman J. Effects of low-dose paroxetine 7.5 mg on weight and sexual function during treatment of vasomotor symptoms associated with menopause. Menopause. 2014 Oct;21(10):1082-90. doi: 10.1097/GME.0000000000000210. PMID 24552977
- [Derived] Simon JA, Portman DJ, Kaunitz AM, Mekonnen H, Kazempour K, Bhaskar S, Lippman J. Low-dose paroxetine 7.5 mg for menopausal vasomotor symptoms: two randomized controlled trials. Menopause. 2013 Oct;20(10):1027-35. doi: 10.1097/GME.0b013e3182a66aa7. PMID 24045678
- See also: Sponsor — http://www.noven.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24-week, multicenter, double-blind, randomized, placebo-controlled study of Brisdelle (paroxetine mesylate) Capsules in subjects with moderate to severe postmenopausal vasomotor symptoms.
  Locations: Medical Clinics
Groups:
- Brisdelle (Paroxetine Mesylate) Capsules: Experimental
  Eligible subjects were randomized to receive either Brisdelle (paroxetine mesylate) Capsules or placebo capsules in a 1:1 ratio.
- Placebo Capsules: Eligible subjects were randomized to receive either Brisdelle (paroxetine mesylate) Capsules or placebo capsules in a 1:1 ratio.
Period: Overall Study
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Started | 285 | 285
Completed | 235 | 218
Not Completed | 50 | 67
Not completed — Adverse Event | 15 | 15
Not completed — Lost to Follow-up | 9 | 3
Not completed — Withdrawal by Subject | 21 | 40
Not completed — Protocol Violation | 1 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Other | 0 | 1
Not completed — Suicidality Tracking Scale | 3 | 1
Not completed — Eligibility Criteria | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules | Total
Number analyzed (Participants) | 285 | 285 | 570
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 269 | 267 | 536
  >=65 years | 16 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (5.47) | 54.5 (5.74) | 54.4 (5.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 285 | 285 | 570
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 285 | 285 | 570

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Hot Flash Frequency at Week 4 and Week 12.
Description: Subjects recorded the number of hot flashes per week using an electronic diary. The results reported are not hot flashes per week.
  The results reported are:
  * Mean Baseline frequency of moderate to severe VMS
  * Mean change in frequency of moderate to severe VMS from baseline to Week 4
  * Mean change in frequency of moderate to severe VMS from baseline to Week 12
Time Frame: Week 4 and Week 12
Population: The outcome data presented for these measurements were obtained using a scale questionnaire. Data were analyzed only from participants who completed and turned in the questionnaire. Therefore, the number of participants analyzed is not consistent with numbers provided in any of the rows in the participant flow module.
Measure: Mean (Standard Deviation); unit: Hot flashes per day
Groups:
- Brisdelle (Paroxetine Mesylate) Capsules; Placebo Capsules: Eligible subjects were randomized to receive either Brisdelle (paroxetine mesylate) Capsules or placebo capsules in a 1:1 ratio.
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Number analyzed (Participants) | 284 | 284
Hot flashes per day
  Baseline | 10.83 (3.86) | 10.90 (3.96)
  Week 4 | -4.13 (4.02) | -2.71 (4.31)
  Week 12 | -5.31 (4.67) | -3.94 (5.13)
Statistical Analysis 1: Comparison: Brisdelle (Paroxetine Mesylate) Capsules vs Placebo Capsules; Test type: Superiority or Other; p < 0.0001, Rank transformed ANCOVA — Week 4 frequency
Statistical Analysis 2: Comparison: Brisdelle (Paroxetine Mesylate) Capsules vs Placebo Capsules; Test type: Superiority or Other; p = 0.0001, Rank transformed ANCOVA — Week 12 frequency

2. Secondary Outcome: Percent Persistence of Benefit, Statistically Significant Difference in Having 50% or More Reduction Compared to Baseline at Week 24.
Description: Persistence of treatment benefit to 24 weeks post treatment was assessed by using the following responder analysis. Responders were defined as those subjects who achieved ≥ 50% reduction from baseline in moderate to severe hot-flash frequency at Week 24; the percent change in hot flash frequency is calculated using the formula:
  Percent reduction at week 24 = [(number of moderate to severe hot flash frequency at baseline - number of moderate to severe hot flash frequency at week 24) / number of moderate to severe hot flash frequency at baseline ]*100%.
Time Frame: Week 24
Population: The outcome data presented for these measurements were obtained using a scale questionnaire. Data were analyzed only from participants who completed and turned in the completed questionnaire. Therefore, the number of participants analyzed is not consistent with numbers provided in any of the rows in the participant flow module.
Measure: Number; unit: percentage of total number of subjects
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Number analyzed (Participants) | 284 | 284
percentage of total number of subjects | 47.54 | 36.27
Statistical Analysis 1: Comparison: Brisdelle (Paroxetine Mesylate) Capsules vs Placebo Capsules; Test type: Superiority or Other; p = 0.0066, Logit model — Week 24 persistence of effect

3. Secondary Outcome: Change in Frequency of Moderate to Severe Hot Flashes Frequency From Baseline (BMI <32 kg/m2, Week 4 and Week 12), Median
Description: Subjects were weighed at each clinic visit and reported the number of hot flashes using an electronic diary.
  For the BMI <32 kg/m2 subgroup, the mean weekly reduction in frequency of moderate to severe hot flashes from Baseline was calculated for Week 4 and Week 12.
Time Frame: Week 4 and Week 12
Population: as for outcome 2
Measure: Median (Full Range); unit: Hot flashes per week
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Number analyzed (Participants) | 197 | 179
Hot flashes per week
  Week 4 | -28.50 [-130 to 48.00] | -18.0 [-151 to 119.0]
  Week 12 | -41.00 [-150 to 119.0] | -27.00 [-168 to 127.0]

4. Secondary Outcome: Change From Baseline in Total Number of Awakenings Due to Hot Flashes, Median
Description: Participants completed a electronic diary to report nightime awakenings. Subjects took study drug once daily at bedtime and they were instructed to complete daily hot flash and sleep diaries to record the number of hot flashes daily, the severity of each episode of hot flash and total number of awakenings due to hot flashes.
  The diary data was used to evaluate and compare the treatment groups, on the change from baseline to Week 4 and Week 12, in the total number of awakenings due to hot flashes. The total number of awakenings due to hot flashes in the run-in period was used as baseline.
Time Frame: Week 4 and Week 12
Population: as for outcome 2
Measure: Median (Full Range); unit: Awakenings
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Number analyzed (Participants) | 255 | 241
Awakenings
  Week 4 | -8.50 [-78.1 to 46.00] | -6.62 [-47.0 to 34.00]
  Week 12 | -13.15 [-80.1 to 49.00] | -8.67 [-47.5 to 22.67]

5. Secondary Outcome: Change in Frequency of Moderate to Severe Hot Flashes Frequency From Baseline (BMI ≥32 kg/m2, Week 4 and Week 12), Median
Description: Subjects were weighed at each clinic visit and reported the number of hot flashes using an electronic diary.
  For the BMI ≥32 kg/m2 subgroup, the mean weekly reduction in frequency of moderate to severe hot flashes from Baseline was calculated for Week 4 and Week 12.
Time Frame: Week 4 and Week 12
Population: as for outcome 2
Measure: Median (Full Range); unit: Hot flashes per week
Groups:
- Brisdelle (Paroxetine Mesylate) Capsules: Eligible subjects were randomized to receive either MesaBrisdelle (paroxetine mesylate) Capsules fem or placebo capsules in a 1:1 ratio.
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Number analyzed (Participants) | 60 | 65
Hot flashes per week
  Week 4 | -22.0 [-118 to 30.00] | -17.0 [-93 to 140.0]
  Week 12 | -31.50 [-124 to 38.00] | -23.00 [-93 to 57.00]

6. Secondary Outcome: Change in Severity of Moderate to Severe Hot Flashes From Baseline (BMI <32 kg/m2, At Week 4 and Week 12), Median
Description: Subjects were weighed at each clinic visit and reported the number of hot flashes using an electronic diary.
  For the BMI <32 kg/m2 subgroup, the mean weekly reduction in the severity of moderate to severe hot flashes from Baseline was calculated at Week 4 and Week 12.
  Subjects recorded the number of hot flashes per week using an electronic diary. Severity score for hot flashes for each subject was calculated as the sum of 2 times the number of moderate hot flashes, plus 3 times the number of severe hot flashes, divided by the total number of moderate and severe hot flashes.
  Weekly Severity Score = (2•Fm +3•FS)/(Fm + FS) Daily Severity Score = {(2•F) m +3•FS)/(Fm + FS)}/7 Where, Fm= Frequency of Moderate Hot Flashes Fs = Frequency of Severe Hot Flashes The calculated severity score is reported below.
Time Frame: Week 4 and Week 12
Population: as for outcome 2
Measure: Median (Full Range); unit: Hot Flash Severity scores per week
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Number analyzed (Participants) | 187 | 173
Hot Flash Severity scores per week
  Week 4 | -0.033 [-1.0 to 0.50] | -0.004 [-1.0 to 0.70]
  Week 12 | -0.045 [-1.0 to 0.89] | -0.00 [-1.0 to 0.74]

7. Secondary Outcome: Change in Severity of Moderate to Severe Hot Flashes From Baseline (BMI ≥32 kg/m2, Week 4 and Week 12), Median
Description: Subjects were weighed at each clinic visit and reported the number of hot flashes using an electronic diary.
  For the BMI ≥32 kg/m2 subgroup, the mean weekly reduction in the severity of moderate to severe hot flashes from Baseline was calculated at Week 4 and Week 12.
  Subjects recorded the number of hot flashes per week using an electronic diary. Severity score for hot flashes for each subject was calculated as the sum of 2 times the number of moderate hot flashes, plus 3 times the number of severe hot flashes, divided by the total number of moderate and severe hot flashes.
  Weekly Severity Score = (2•Fm +3•FS)/(Fm + FS) Daily Severity Score = {(2•F) m +3•FS)/(Fm + FS)}/7 Where, Fm= Frequency of Moderate Hot Flashes Fs = Frequency of Severe Hot Flashes The calculated severity score is reported below.
Time Frame: Week 4 and Week 12
Population: as for outcome 2
Measure: Median (Full Range); unit: Hot Flash Severity scores per week
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Number analyzed (Participants) | 58 | 63
Hot Flash Severity scores per week
  Week 4 | -0.039 [-0.94 to 0.81] | -0.036 [-0.56 to 0.71]
  Week 12 | -0.052 [-0.57 to 0.97] | -0.051 [-1.0 to 0.71]

8. Secondary Outcome: Change From Baseline in Greene Climacteric Scale (GCS) at Week 4 and Week 12, Total Score, Median
Description: The Greene Climacteric Scale (GCS) was used for this measurement. The scale has 21 questions and measures symptoms in 4 areas; these are psychological (anxiety and depression), physical, vasomotor, and libido.
  The severity of the symptom was scored as: 0=none, 1=mild, 2=moderate, and 3=severe. Anxiety was determined by using the sum of scores 1 to 6, and depression was determined by using the sum of scores 7 to 11. Physical aspects were determined by using the sum of scores 12 to 18; vasomotor aspects were determined by using the sum of scores 19 to 20; and libido was determined by using the score for question 21.
  The total GCS score ranges from "0" to "63" which is the sum of all the scores for the 21-symptom assessment questions in this scale. Each subject's total GCS score at baseline and at Week 4 and Week 12 were used to calculate change from baseline in these symptoms. The change from baseline is reported below.
Time Frame: Week 4 and Week 12
Population: as for outcome 2
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Number analyzed (Participants) | 216 | 203
units on a scale
  Week 4 | -3.00 [-36 to 16.00] | -3.00 [-37 to 13.00]
  Week 12 | -4.00 [-33 to 14.00] | -3.00 [-32 to 48.00]

9. Secondary Outcome: Percentage of Responders
Description: Participants reported the number of hot flashes using an electronic diary. Participants who hd a ≥50% reduction in hot flash frequency were defined as responders. The percent of responders is presented below.
Time Frame: Week 4 and Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Number analyzed (Participants) | 284 | 284
percentage of participants
  Week 4 | 35.56 | 25.35
  Week 12 | 49.30 | 33.80

10. Secondary Outcome: Percent Daytime and Nighttime Responders, Numerical Rating Scale (NRS)
Description: Subject's overall improvement in VMS from Baseline assessed using the Numerical Rating Scale (NRS) The NRS is measured on a scale of 0 to 10 on how bothered the subject was by her VMS (0=not bothered at all and 10=very much bothered).
  Responders: Subjects with NRS Score of 5 Or Less. Non-Responders: Subjects With NRS Score of Greater than Or Equal to 6.
Time Frame: Week 4 and Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of total number of subjects
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Number analyzed (Participants) | 281 | 281
percentage of total number of subjects
  Week 4 | 35.48 | 25.27
  Week 12 | 46.62 | 37.72

11. Secondary Outcome: Change From Baseline in Arizona Sexual Experience Scale (ASEX, Week 4 and Week 12) Total Score, Median
Description: The Arizona Sexual Experiences Scale (ASEX) is a 5-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm. Possible total scores range from 5 to 30, with the higher scores indicating more sexual dysfunction.The sum of the scores for all 5 items was calculated at Week 4 and Week 12.
Time Frame: Week 4 and Week 12
Population: as for outcome 2
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Number analyzed (Participants) | 202 | 216
Units on a scale
  Week 4 | 0.00 [-3.00 to 4.00] | 0.00 [-3.00 to 4.00]
  Week 12 | 0.00 [-3.00 to 4.00] | 0.00 [-3.00 to 3.00]

12. Secondary Outcome: Effect of Paroxetine Mesylate Capsules on Percent Improvement of Hot Flash Interference From Baseline at Week 4 and Week 12, Hot Flash Related Daily Interference Scale (HFRDIS)
Description: Interference of hot flashes was measured by using the hot flash-related daily interference scale (HFRDIS). The HFRDIS is a 10-item scale that measures the degree to which hot flashes interfere with 9 daily activities and the tenth item measures the degree to which hot flashes interfere with each of the other items. Subjects can score for each item on a scale from 0 to 10 where 0 = Do not interfere and a score of 10 = Completely interferes.
  The measure being reported below is percentage of responders who had an improvement in HFRDIS score at Week 4 and Week 12 compared to baseline. A responder is defined as a subject who had an improvement in the HFRDIS score. An improvement is defined as a score ≤3 on each question.
Time Frame: Week 4 and Week 12
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Number analyzed (Participants) | 214 | 197
Percent of participants
  Week 4 | 26.03 | 30.51
  Week 12 | 15.89 | 21.32

13. Secondary Outcome: Percent Responders Improvement in VMS From Baseline Using the Clinical Global Impression (CGI) Scale.
Description: Proportion of NRS Responders: Subject's overall improvement in VMS from Baseline was assessed using the Numerical Rating Scale (NRS)
  The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  Responders: Subjects Achieving a Score of "Very Much Improved" Or "Much Improved" Or "Minimally Improved".
  Non Responders: Subjects with a Score of "No Change" Or "Minimally Worse" Or "Much Worse" Or "Very Much Worse".
Time Frame: Week 4 and Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Number analyzed (Participants) | 249 | 231
percentage of participants
  Week 4 | 67.88 | 53.58
  Week 12 | 69.88 | 59.74

14. Secondary Outcome: Effect of Brisdelle (Paroxetine Mesylate) Capsules on Anxiety and Depression
Description: Depression & anxiety were measured by using the Hospital Anxiety & Depression Scale (HADS).
  The HADS was developed to assess anxiety & depression. It is meant to differentiate symptoms of depression with those of anxiety.
  Number of items: 14 (7 questions relating to anxiety; 7 questions relating to depression).
  Responses are based on the relative frequency of symptoms over the past week, using a four point scale ranging from 0 (not at all) to 3 (very often indeed).
  Responses are summed to provide separate scores for anxiety and depression symptomology with possible scores ranging from 0 to 21 for each scale.
  The results presented below are the percentage of participants with abnormal HADS Scores for both Abnormal Anxiety & Abnormal Depression at Week 4 and Week 12.
Time Frame: Week 4 and Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Number analyzed (Participants) | 218 | 210
Percentage of participants
  Week 4 | 5.65 | 2.44
  Week 12 | 4.13 | 5.24

15. Secondary Outcome: Assessment of Mood
Description: Mood was measured by using the Profile of Mood States (POMS) questionnaire. The Profile of Moods States (POMS) is a 65-item multi-dimensional measure that provides a method of assessing transient, fluctuating active mood states. Key areas that are measured include: tension-anxiety, anger-hostility, fatigue-inertia, depression-dejection, vigor-activity, confusion-bewilderment. Responses to questions are scored with the following numerical values: Not at all = 1, A little = 2, Moderate = 3, Quite a bit = 4, Extremely = 5. A total score for a domain was obtained by summing the responses of individual items in the domain. The total POMS score can range from "65" to "325." Each subject's total POMS score at baseline and at Week 4 and Week 12 were used to calculate the percent of participants with less disturbance in mood at Week 4 and Week 12 compared to baseline. The percent of participants with less disturbance in mood is reported below.
Time Frame: Week 4 and Week 12
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Number analyzed (Participants) | 218 | 208
Percent of participants
  Week 4 | 37.40 | 42.39
  Week 12 | 37.16 | 44.23

16. Secondary Outcome: BMI Change From Baseline (kg/m2), Median
Description: Subjects were weighed at each clinic visit and reported the number of hot flashes using an electronic diary.
  Assessment of the effect of Brisdelle compared with placebo on body mass index.
Time Frame: Week 4 and Week 12
Population: as for outcome 2
Measure: Median (Full Range); unit: kg/m2
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Number analyzed (Participants) | 250 | 233
kg/m2
  Week 4 | 0.00 [-2.17 to 2.66] | 0.08 [-3.08 to 9.15]
  Week 12 | 0.15 [-2.33 to 2.10] | 0.11 [-2.56 to 9.70]

17. Primary Outcome: Mean Change From Baseline in Hot Flash Severity at Week 4 and Week 12.
Description: Subjects recorded the number of hot flashes per week using an electronic diary. Severity score for hot flashes for each subject was calculated as the sum of 2 times the number of moderate hot flashes, plus 3 times the number of severe hot flashes, divided by the total number of moderate and severe hot flashes.
  Weekly Severity Score = (2•Fm +3•FS)/(Fm + FS) Daily Severity Score = {(2•F) m +3•FS)/(Fm + FS)}/7 Where, Fm= Frequency of Moderate Hot Flashes Fs = Frequency of Severe Hot Flashes
Time Frame: Week 4 and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hot Flash Severity Score per day
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Number analyzed (Participants) | 284 | 284
Hot Flash Severity Score per day
  Baseline | 2.525 (0.30) | 2.532 (0.32)
  Week 4 | -0.092 (0.24) | -0.059 (0.22)
  Week 12 | -0.0126 (0.31) | -0.066 (0.26)
Statistical Analysis 1: Comparison: Brisdelle (Paroxetine Mesylate) Capsules vs Placebo Capsules; Test type: Superiority or Other; p = 0.0368, Rank transformed ANCOVA — Week 4 severity
Statistical Analysis 2: Comparison: Brisdelle (Paroxetine Mesylate) Capsules vs Placebo Capsules; Test type: Superiority or Other; p = 0.0064, Rank transformed ANCOVA — Week 12 severity

ADVERSE EVENTS:
Time Frame: 24 Weeks
Arm/Group | Brisdelle (Paroxetine Mesylate) Capsules | Placebo Capsules
Serious Adverse Events (participants affected / at risk) | 13/285 | 7/285
Other Adverse Events (participants affected / at risk) | 161/285 | 146/285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brisdelle (Paroxetine Mesylate) Capsules (N=285) | Placebo Capsules (N=285)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 3 (3) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brisdelle (Paroxetine Mesylate) Capsules (N=285) | Placebo Capsules (N=285)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (3) | 0 (0)
Eye allergy (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Retinal degeneration (Eye disorders) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 2 (2)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 9 (10)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 4 (4)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (2) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 13 (14) | 3 (3)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sensitivity of teeth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 3 (3) | 1 (1)
Cyst (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 12 (12) | 7 (7)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Feeling jittery (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 2 (2) | 6 (6)
Malaise (General disorders) | 1 (1) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 3 (3) | 1 (1)
Pain (General disorders) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 8 (8) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 3 (3) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 4 (4) | 7 (7)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 9 (10) | 7 (7)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 20 (20) | 20 (22)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 2 (2) | 0 (0)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 15 (16) | 13 (14)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (2)
Tooth abscess (Infections and infestations) | 2 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 12 (15) | 18 (20)
Urinary tract infection (Infections and infestations) | 4 (4) | 3 (3)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Sciatic nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood glucose abnormal (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 3 (3) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 5 (5)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1)
Heart rate irregular (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 2 (2)
Vitamin D decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Weight increased (Investigations) | 2 (2) | 3 (3)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Circadian rhythm sleep disorder (Nervous system disorders) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 3 (3)
Dysgeusia (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 12 (12) | 8 (11)
Hyperreflexia (Nervous system disorders) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 4 (4) | 0 (0)
Lethargy (Nervous system disorders) | 2 (2) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 4 (4) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Serotonin syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 2 (2)
Abnormal dreams (Psychiatric disorders) | 3 (3) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 2 (2)
Anger (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (3) | 7 (9)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 4 (4)
Elevated mood (Psychiatric disorders) | 0 (0) | 1 (1)
Emotional disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 8 (8)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1)
Loss of libido (Psychiatric disorders) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 4 (4) | 3 (3)
Nervousness (Psychiatric disorders) | 1 (2) | 1 (1)
Nightmare (Psychiatric disorders) | 2 (2) | 2 (2)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 2 (3)
Self esteem decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 4 (4) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Tearfulness (Psychiatric disorders) | 1 (1) | 0 (0)
Thinking abnormal (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (3) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 1 (3)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Sexual dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 (4) | 2 (2)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 2 (2)
Sweat gland disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dental operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Meniscus operation (Surgical and medical procedures) | 1 (1) | 1 (1)
Sinus operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other